CLINICAL TRIAL: NCT01434108
Title: Effects of the Administration of Ornithine Phenylacetate in Patients With Cirrhosis and Upper Gastrointestinal Bleeding
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OP_GIB; 2009-017819-16 (EudraCT Number)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Bleeding; Cirrhosis
Keywords: cirrhosis, gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Fibrosis | interventions — ornithine phenylacetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ornithine-phenylacetate (Experimental): Administration of OP (OCR-002) during 5 days in addition to standard treatment of gastrointestinal bleeding.
  Interventions: Drug: Ornithine-phenylacetate
- Saline iv (Placebo Comparator): Administration of control infusion (saline infusion) during 5 days in addition to standard treatment of gastrointestinal bleeding.
  Interventions: Drug: Ornithine-phenylacetate

INTERVENTIONS:
Drug: Ornithine-phenylacetate — Phase A: Open-label scalating dose of OP. Treatment will be initiated at 1/3 of the final dose and will be scalated every 12 hours up to the full dose, except if there are problems of tolerance. Duration of the infusion 5 days.
  Phase B: Comparative study of experimental drug vs placebo for 5 days OP (OCR-002) at a dose of 10 g diluted in 150 ml of water for injection administered as a continuous i.v. infusion for 24 hours (8.3 ml/h)during 5 days.
  Other Names: OCR-002

SUMMARY:
The main objective is to evaluate the effectiveness of the experimental drug to reduce plasma ammonia concentration at a dose that is safe and well tolerated. Ammonia usually rises significantly in the hours after gastrointestinal bleeding in patients with cirrhosis of the liver. This increase in the concentration of ammonia facilitates the development of hepatic encephalopathy.

The study will be divided in two parts:

Part A: Open-label, dose-escalating, single cohort study. The goal of this phase is to confirm the tolerance and safety of the dose of OP that is being proposed for the study according to the results of phase I and phase II studies in healthy subjects and stable outpatients with cirrhosis.

Part B: Multi-center (2 University Hospitals), double-blind, randomized, parallel-group trial. Assignment of treatment will be done according to a list (one at each study site) of random numbers in blocks that will be concealed until the end of the study. The control group will be assigned to placebo on a 1:1 ratio. The placebo and treatment will be masked.

ELIGIBILITY:
Inclusion criteria

* Cirrhosis of the liver; diagnosed by clinical, laboratory or radiological findings.
* Upper gastrointestinal bleeding, as judged by clinical signs (hematemesis, melena, anemia) combined with endoscopic data.
* Bleeding that has been active within 24 hours prior to inclusion; signs of activity are defined by the presence of blood in the gastrointestinal tract and symptoms attributable to bleeding (hypotension, tachycardia, etc.).
* Age between 18 and 75 years.
* Informed consent by the patient. In case of inability to provide informed consent due to impaired mental status secondary to hepatic encephalopathy the informed consent should be provided by the next of kin and should be confirmed by the patient when he/she recovers from hepatic encephalopathy.
* Absence of exclusion criteria.

Exclusion criteria

* Terminal illness (e.g. advanced hepatocellular carcinoma).
* Need for mechanical ventilation.
* Renal impairment, defined by a creatinine > 1.5 mg/dl or need of hemodialysis.
* Pregnant or breast-feeding. Pre-menopausal women capable of bearing children should be following a reliable method of birth control and should have a negative result in a pregnancy test prior to inclusion.
* Known or suspected hypersensitivity or allergic reaction to ornithine or phenylacetate.
* Use of medications known to interfere with the clearance of either ornithine and/or phenylacetate, such as antibiotics of the penicillin group and probenicid.
* Use of medications that may induce hyperammonemia; such as haloperidol, valproic acid, and systemic corticosteroids.
* History or known infection with human immunodeficiency virus (HIV).
* Neurological comorbidities that impair mental status and do not allow to adequately assess the presence or outcome of hepatic encephalopathy.
* The presence in the electrocardiogram of a QTcF >500 msec

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Ammonia plasma concentration umol/L. | 6 days
  Venous plasma ammonia will be assessed within 60 minutes of extraction in samples withdrawn every 12 hours during the first 48 hours and once a day during the second 72 hours. The concentration of ammonia will be used to decide: a)dose escalating in the initial phase (first 48 hours) of part A and b)discontinuation of treatment in the second phase (second 72 hours) of part B. Blood samples will be processed immediately after being withdrawn to separate plasma under cold conditions. Ammonia will be measured enzymatically in a Cobas Integra analyzer.

SECONDARY OUTCOMES:
Hepatic encephalopathy | 6 days
  Hepatic encephalopathy (HE) is a common complication of cirrhosis,characterized by a myriad of neurological manifestations,diverse underlying liver disorders, and a variety of precipitating factors. For evaluated the presence and severity of HE the CHESS, and WEST-HAVEN scales will be performe because are adequate for clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Genescà, MD, Principal Investigator — EASL
Locations (1):
- Hospital Vall Hebron, Barcelona, Barcelona, Spain